CLINICAL TRIAL: NCT02872727
Title: Nanoparticles Emitted by Aircraft Engines, Impact on the Respiratory Function: Cohort Follow-up Study
Brief Title: Nanoparticles Emitted by Aircraft Engines, Impact on the Respiratory Function:
Acronym: NANOAF2
Status: Terminated | Type: Observational
Why Stopped: Inclusion of the last patient
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Aix Marseille Université (Other); LBM- Nanosecurity platform - CEA Grenoble (Unknown); LR2N - Nanosecurity platform - CEA Grenoble (Unknown)
Responsible Party: Sponsor
Other Study IDs: 9637; 2015-A01771-48 (Other: RCB number)
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Air France Company's Employees Working in the Marseilles and Paris Airports (Flightline and Administrative Employees)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Exhaled air and urine samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Air France Company's Employees Working: Observational cohort : Air France Company's Employees Working in the Marseilles and Paris Airports having Respiratoy health, biological investigations
  Interventions: Other: Respiratoy health, biological investigations

INTERVENTIONS:
Other: Respiratoy health, biological investigations — Once the subjects have agreed to participate, self-surveys on their lifestyle habits will be filled and EACand urine samplings will be taken during one same consultation, in addition to exhaled CO and No measurements. This consultation will also include a spirometry test. The employees' workstation data (and their evolution since the first study) will be collected. Therefore, the volunteers' participation is limited to one single visit including non-invasive examinations and self-surveys.

SUMMARY:
The object of this new project is to proceed with investigations with the employees of the cohort for the first study so as to obtain a remote evolution (5 years) of their respiratory function while measuring their nanoparticle exposure. This will enable us to assess the possible link between exposure and respiratory function evolution in the employees

DETAILED DESCRIPTION:
It is well known that the nanoparticle (NP) rate is higher in large metropolitan cities but also in the airport environments owing to aircraft engine emissions. Now, this nanoparticulatepollution is a public health issue owing to its potential cardiovascular and respiratory impact on general population. Besides, an evolution of exposure in airport environments is now observed, due to the implementation of new protective equipment better adapted to nanoparticles and to the use of new fuels.

From October 2011 to June 2012, our partnership network conducted a first study on the assessment of the respiratory health of the Air France company'semployees working in the Marseillesand Paris airports (flightline and administrative employees). This study was promoted by the Montpellier CHRU, Regional University Hospital Centre (ANSM identification number 2011-A00646-35). It allowed 471 voluntary employees to be involved. They answered a lifestyle survey and underwent a spirometry, an exhaled CO measurement and a sampling of exhaled air condensate (EAC). A metrological study of particles emitted by aircraft engines and found in the airport environment was conducted and the elementary chemical composition analysis, as well a sieve analysis of particles present in the EACwere conducted. The data analysis from this first study (whose publications are currently being drafted) gave rise to a description of the respiratory health condition of the employees working in the vicinity of nanoparticle production sources, and to characterise exposure to nanoparticles of secondary emission originating from aircraft engine exhaust gases, as well as a description of the elementary and particulate content of the EACsin this whole population.

The analysis of the respiratory functions of the exposed subjects combined with the measurement and characterisation of nanoparticlesemitted by aircraft engines (through a metrology data analysis) and with the EACanalysis allowed the measurement of the exposure levels and the assessment of the respiratory health of the employees in an airport environment. Besides, the studied population was located on two airports in two different cities (Roissy Charles de Gaulle for Paris and Marignanefor Marseilles).

So far, no longitudinal follow-up study of airport NPsin a large size sample has been carried out, notably in a plurisdisciplinary scope. Yet only such a longitudinal follow-up analysis of the cohortwill provide a suitable impact study of the various exposure factors, taking into account their integration. Now, no large size cohortof subjects exposed to secondary emission nanoparticlesor ultrafine particles (UFP) has ever been monitored in France.

The first previously conducted study enabled us to draw up a situational respiratory health analysis on 471 employees. It also allowed us to measure nanoparticlesin their exhaled air and to evaluate their UFPexposure rate on the work station. It is now relevant to monitor the evolution of these parameters in the course of time and better assess the role of possibly confounding factors in the evolution of their respiratory health.

The EAC is collected by means of a simple device and is a non-invasive tool providing useful information on lung exposure, or even on inflammatory effects at respiratory tract level. The EACis a good proposed methodology to study exposure and effect biomarkers in professional exposure situations (Mutti 2006; Corradi 2010). Exposure biomarkers such as metals were also studied in the EACin connection with smoking (Mutti 2006) or with professional exposure to metallic particles (Goldoni 2010, Goldoni2004, Hoffmeyer2011). In a recent study, the EACwas used in order to locate nanoparticlesand oxidative stress markers (malondialdehydeand hydrogen peroxide H2O2) in volunteers exposed to cigarette smoke (Sauvain 2014). As the EACis a highly diluted aqueous medium, there is no reported matrix effect. However, one of the difficulties lies in the use of highly sensitive techniques. In the scope of our previous study, the analysis techniques were already implemented and used on the 471 collected EACsamples. The Medical Biology Laboratory of CEA in Grenoble is currently working on methodologies intended to standardise the analyses in this medium (sodium measured in parallel by ICPMS, knowing that standardisation was proposed in the literature: Dompeling 2010) and other methodologies such as total protein assaying by µBCA.

The object of this new project is to proceed with investigations with the employees of the cohort for the first study so as to obtain a remote evolution (5 years) of their respiratory function while measuring their nanoparticle exposure. This will enable us to assess the possible link between exposure and respiratory function evolution in the employees

ELIGIBILITY:
Inclusion Criteria:

* Subject must be given free and informed consent and signed the consent
* Subject must be affiliated or beneficiary in a health insurance plan
* Subject included in our previous study (RBC No: 2011-A00646-35; NCT03098784)

Exclusion Criteria:

- Subject has a cons-indication (or an incompatible combination therapy) for the realization of the EFR.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects previously included in our previous study (RBC No: 2011-A00646-35; NCT03098784).
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2020-12-13 (Actual); Study Completion 2021-06-13 (Actual)

PRIMARY OUTCOMES:
respiratory function | 1 day (Day of inclusion (D0))
  maximum expiratory volume per second (MEVS)

SECONDARY OUTCOMES:
Exhaled CO measurement | 1 day (Day of inclusion (D0))
  Exhaled CO measurement
Exhaled NO measurement | 1 day (Day of inclusion (D0))
  Exhaled NO measurement
Exhaled air condensate | 1 day (Day of inclusion (D0))
  Exhaled air condensate
oxidative stress marker (8 isoprostane) | 1 day (Day of inclusion (D0))
  oxidative stress marker (8 isoprostane)
plasma mass spectrometry which allows the simultaneous assaying of 17 elements | 1 day (Day of inclusion (D0))
  plasma mass spectrometry which allows the simultaneous assaying of 17 elements (Zn, Al, Ti, Co, Cu, Zr, Ni, Cr, Ga, In, Mn, Fe, Se, Cd, Ge, Be)

CONTACTS AND LOCATIONS:
Overall Officials: NICOLAS MOLINARI, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided